CLINICAL TRIAL: NCT03378934
Title: A Single-center, Randomized, Open-label, Controlled, Dose-escalating, Parallel-group Study to Assess the Anti-platelet Effect of Berberine in Patients Receiving Aspirin and Clopidogrel After Percutaneous Coronary Intervention
Brief Title: Anti-platelet Effect of Berberine in Patients After Percutaneous Coronary Intervention
Acronym: APLABE-PCI
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, LiuZhenyu, Professor, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-I2M-1-011; JS-1375 (Other: Ethics Committee in Peking Union Medical College Hospital)
Record Dates: First submitted 2017-12-14; First posted 2017-12-20 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Coronary Artery Disease; Percutaneous Coronary Intervention
Keywords: Coronary Artery Disease; Percutaneous Coronary Intervention; Antiplatelet; Berberine
MeSH Terms: conditions — Coronary Artery Disease | interventions — Berberine; Aspirin; Clopidogrel

STUDY DESIGN:
Intervention Model Description: On the first day of the treatment period (Visit 1), eligible patients will be randomized into the Berberine Arm and the Control Arm.
  In the Berberine Arm, patients will receive berberine 200 mg twice daily for 4±1 weeks (Stage 1); then, 300 mg twice daily for 4±1 weeks (Stage 2); then, 400 mg twice daily for 4±1 weeks (Stage 3) in addition to standard treatment, including aspirin 100 mg once daily and clopidogrel 75 mg once daily for 12±1 weeks.
  In the Control Arm, patients will receive standard treatment, including aspirin 100 mg once daily and clopidogrel 75 mg once daily for 12±1 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Berberine Arm (Experimental): In the Berberine Arm, patients will receive berberine 200 mg twice daily for 4±1 weeks (Stage 1); then, 300 mg twice daily for 4±1 weeks (Stage 2); then, 400 mg twice daily for 4±1 weeks (Stage 3) in addition to standard treatment, including aspirin 100 mg once daily and clopidogrel 75 mg once daily for 12±1 weeks.
  Interventions: Drug: Berberine; Drug: Standard treatment; Drug: Aspirin; Drug: Clopidogrel
- Control Arm (Active Comparator): In the Control Arm, patients will receive standard treatment, including aspirin 100 mg once daily and clopidogrel 75 mg once daily for 12±1 weeks.
  Interventions: Drug: Standard treatment; Drug: Aspirin; Drug: Clopidogrel

INTERVENTIONS:
Drug: Berberine — Berberine 200 mg twice daily for 4±1 weeks (Stage 1); then, 300 mg twice daily for 4±1 weeks (Stage 2); then, 400 mg twice daily for 4 weeks (Stage 3).
  Other Names: Berberine Hydrochloride Tablets
  Arms: Berberine Arm
Drug: Standard treatment — Standard treatment for 12±1 weeks.
Drug: Aspirin — Aspirin 100 mg once daily for 12±1 weeks.
  Other Names: Aspirin Enteric-coated Tablets; Bayaspirin
Drug: Clopidogrel — Clopidogrel 75 mg once daily for 12±1 weeks.
  Other Names: Clopidogrel Hydrogen Sulphate Tablets; Plavix

SUMMARY:
The APLABE-PCI is a single-center, randomized, open-label, controlled, dose-escalating, parallel-group study, which is designed to assess the anti-platelet effect of berberine in approximately 64 patients receiving aspirin and clopidogrel who are at > 8 but ≤ 40 weeks after percutaneous coronary intervention.

DETAILED DESCRIPTION:
Background

Dual antiplatelet therapy (DAPT) with aspirin and a platelet P2Y12 inhibitor is mandatory in patients after percutaneous coronary intervention (PCI). Clopidogrel is the most widely used P2Y12 inhibitor with class I recommendation. However, clopidogrel is a pro-drug which has highly variable antiplatelet effect. Hypo-responsiveness to clopidogrel was associated with increased risk of thrombotic events after PCI.

Increasing the dose of aspirin could not reduce thrombotic risk but resulted in elevated bleeding risk. Although new P2Y12 inhibitors have more potent antiplatelet effect and did reduce thrombotic risk compared with clopidogrel, the benefit was only demonstrated in patients undergoing PCI for moderate to high risk non-ST-segment elevation acute coronary syndrome (NSTE-ACS) or ST-segment elevation myocardial infarction (STEMI) and was also associated with increased bleeding risk. Therefore, how to improve the antiplatelet therapy in patients taking aspirin and clopidogrel after PCI remains unclear.

Berberine is an isoquinoline plant alkaloid which has anti-inflammatory, anti-oxidant, anti-microbial, anti-tumoral and immunomodulatory properties, as well as anti-hypertensive, hypo-glycemic and cholesterol-lowering effects. In small studies conducted in patients with hypertension, hypercholesterolemia and diabetes, berberine with a daily dose of 600-1000 mg for 12 weeks had good safety profile and was well tolerated.

In addition, berberine demonstrated antiplatelet effect. After in vivo administration in animals, berberine inhibited ex vivo platelet activation mediated by P2Y12 receptor and ex vivo platelet aggregation induced by adenosine diphosphate (ADP), arachidonic acid (AA), collagen, and thrombin, et al. After ex vivo administration, berberine inhibited ex vivo thromboxane B2 (TXB2) synthesis induced by ADP, AA, and collagen in animal platelets, as well as ex vivo platelet aggregation induced by collagen in a dose-dependent manner in platelets from healthy human volunteers. However, the antiplatelet effect of berberine has never been investigated in patients receiving DAPT after PCI.

Design

The APLABE-PCI is a single-center, randomized, open-label, controlled, dose-escalating, parallel-group study, which is designed to assess the anti-platelet effect of berberine in approximately 64 patients receiving aspirin and clopidogrel who are at > 8 but ≤ 40 weeks after PCI.

The total study duration is expected to be approximately 19 weeks per patient, including a screening period, a 12±1 week treatment period, and a 4±1 week follow-up period.

The visit schedule will be as follows:

* Visit 0 (V0): Day -21 to Day -1, Screening/Enrolment;
* Visit 1 (V1): Day 1, Randomization/First dose;
* Visit 2 (V2): Week 4±1, Dose adjustment 1;
* Visit 3 (V3): Week 8±1, Dose adjustment 2;
* Visit 4 (V4): Week 12±1, End of Treatment (EOT) /Last dose; •Visit 5 (V5): Week 16±1, Safety visit.

The screening period will be up to 21 days. Once each patient has signed the informed consent, the eligibility of the patient will be evaluated and related laboratory assessments will be taken (Visit 0). All patients will continue taking aspirin and clopidogrel in the morning during the screening period.

On the first day of the treatment period (Visit 1), eligible patients will return to the study center and be randomized into the Berberine Arm and the Control Arm. In the Berberine Arm, patients will receive berberine 200 mg twice daily for 4±1 weeks (Stage 1); then, 300 mg twice daily for 4±1 weeks (Stage 2); then, 400 mg twice daily for 4±1 weeks (Stage 3) in addition to standard treatment, including aspirin and clopidogrel. In the Control Arm, patients will receive standard treatment, including aspirin and clopidogrel, for 12±1 weeks. During the treatment period, patients in both arms will also take aspirin 100 mg once daily and clopidogrel 75 mg once daily for 12±1 weeks.

The total daily dose of berberine will be taken separately in the morning and in the evening in approximately a 12-hour interval. On the first day of the treatment period (Visit 1), the morning dose (first dose) of berberine will be given 2-4 hour after aspirin and clopidogrel are taken together in the morning and immediately after the blood and urine samples for baseline platelet function tests are collected. Since the second day of the treatment period, the morning dose of berberine will be taken simultaneously with aspirin and clopidogrel in the morning.

At the ends of Stage 1 (Visit 2), Stage 2 (Visit 3), and Stage 3 (Visit 4) (end of treatment, EOT), patients will return to the study center. During each stage, the last morning doses of all antiplatelet agents, including berberine, aspirin, and clopidogrel in the Berberine Arm, as well as aspirin and clopidogrel in the Control Arm, will be administered simultaneously at the study center in the morning on Visit 2, Visit 3, and Visit 4, respectively.

A follow-up period will begin on the next day after Visit 4 and will continue for 4±1 weeks. During the follow-up period, patients in both arms will continue taking aspirin and clopidogrel. At the end of the follow-up period, patients will return to the study center for a safety visit (Visit 5).

In the Berberine Arm, the blood and urine samples for platelet function tests will be obtained 2-4 hour after aspirin and clopidogrel are taken in the morning and before the first morning dose of berberine is taken on Visit 1, and 2-4 hours after the morning doses of berberine, aspirin and clopidogrel are taken on Visit 2, Visit 3, and Visit 4, respectively. In the Control Arm, the blood and urine samples for platelet function tests will be collected 2-4 hours after the morning doses of aspirin and clopidogrel are given on Visit 1, Visit 2, Visit 3, and Visit 4, respectively.

In the Berberine Arm, the blood and urine samples for safety assessment will be collected on Visit 0, and 2-4 hours after the morning doses of berberine, aspirin and clopidogrel are taken on Visit 2, Visit 3, and Visit 4, as well as on Visit 5, respectively. In the Control Arm, the blood and urine samples for safety assessment will be collected on Visit 0, and 2-4 hours after the morning doses of aspirin and clopidogrel are taken on Visit 2, Visit 3, and Visit 4, as well as on Visit 5, respectively.

Adverse events will be collected on Visit 1, Visit 2, Visit 3, Visit 4, and Visit 5, respectively. Cardiac ischemic events and bleeding events will be collected on Visit 2, Visit 3, and Visit 4, respectively.

The primary endpoint of the study is P2Y12 reaction unit (PRU) assessed by VerifyNow assay 2-4 h after all the antiplatelet agents are taken simultaneously in the morning at the end of the treatment period (Visit 4, EOT), i.e., on the 12th (11th-13th) week of treatment.

Conclusions

The APLABE-PCI study will assess the anti-platelet effect of berberine in patients receiving aspirin and clopidogrel after PCI. The result of the present study would provide pharmacodynamical data for the design of future outcome studies.

ELIGIBILITY:
Inclusion criteria

1. Provision of written informed consent.
2. Aged 18-70 years, male or female.
3. Currently, > 8 but ≤ 40 weeks after index percutaneous coronary intervention (PCI) .
4. Receiving dual antiplatelet therapy (DAPT) with aspirin (Bayaspirin TM) 100 mg once daily and clopidogrel (Plavix TM) 75 mg once daily for ≥ 7 days.
5. No cardiac ischemic events or bleeding events occurred after the index PCI.

   * Cardiac ischemic events include myocardial infarction, coronary revascularization, and definite or probable stent thrombosis;
   * Bleeding events include major or minor bleeding according to the Platelet Inhibition and Patient Outcomes (PLATO) definition.
6. PRECISE-DAPT score < 25 evaluated after the index PCI and before the index hospital discharge.
7. Females who are either post-menopausal > 1 year or surgically sterile.

Exclusion criteria

1. Use of berberine within 30 days of screening.
2. Use of any fibrinolytic or antithrombotic agents, with the exception of aspirin and clopidogrel, within 30 days of screening.
3. Any indications other than coronary artery disease (e.g., atrial fibrillation, prosthetic heart valve, venous thromboembolism, ventricular thrombosis, et al) for fibrinolytic or antithrombotic treatment during the study period.
4. Planned use of berberine, as well as any fibrinolytic or antithrombotic agents, with the exception of aspirin (Bayaspirin TM) and clopidogrel (Plavix TM), during the study period.
5. Planned use of moderate or strong cytochrome P450 (CYP) 2C19 inhibitors, CYP2C19 substrates with narrow therapeutic index, or strong CYP2C19 inducers during the study period.
6. Planned coronary revascularization, including PCI and coronary artery bypass graft (CABG) during the study period.
7. Increased bleeding risk, including

   * any history of intracranial, intraocular, retroperitoneal, or spinal bleeding;
   * recent (within 30 days of screening) gastrointestinal (GI) bleeding;
   * recent (within 30 days of screening) major trauma or major surgery;
   * planned surgery or other invasive procedure during the study period;
   * sustained uncontrolled hypertension (systolic blood pressure [SBP] > 180 mmHg or diastolic blood pressure [DBP] > 100 mmHg);
   * history of hemorrhagic disorders, e.g., haemophilia, von Willebrand's disease;
   * inability to discontinue non-steroidal anti-inflammatory drugs (NSAIDs) during the study period;
   * platelet count less than 100,000/mm3 or hemoglobin < 10 g/dL.
8. Contraindications for aspirin, clopidogrel, and berberine, e.g., hypersensitivity, active bleeding, bleeding diathesis, coagulation disorders, severe liver or kidney diseases, hemolytic anemia, glucose-6-phosphate dehydrogenase deficiency, et al.
9. History of intolerance to aspirin, clopidogrel, and berberine.
10. Any condition, which in the opinion of the Investigator, would make it unsuitable for the patient to participate in this study. For example, conditions which may put the patient at risk, e.g., liver or kidney dysfunction, et al; or increase the risk of non-compliance to study protocol or follow-up, e.g., history of drug addiction or alcohol abuse, et al; or influence the result of the study, e.g., active cancer, et al.
11. Patients who has previously been randomized in this study.
12. Participation in another investigational drug or device study within 30 days of screening.
13. Involvement in the planning and conduct of the study (applies to investigators, contract research organization staff, and study site staff, et al).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2018-09-26 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
P2Y12 reaction unit (PRU) | On the 12th (11th-13th) week of treatment
  The P2Y12 reaction unit (PRU) assessed by VerifyNow assay 2-4 h after all the antiplatelet agents are taken simultaneously in the morning at the end of the treatment period (Visit 4, EOT), i.e., on the 12th (11th-13th) week of treatment

SECONDARY OUTCOMES:
P2Y12 reaction unit (PRU) | On the 8th (7th-9th) week of treatment
  The P2Y12 reaction unit (PRU) assessed by VerifyNow assay 2-4 h after all the antiplatelet agents are taken simultaneously in the morning at the end of Stage 2 (Visit 3) [ i.e., on the 8th (7th-9th) week of treatment ]
P2Y12 reaction unit (PRU) | On the 4th (3rd-5th) week of treatment
  The P2Y12 reaction unit (PRU) assessed by VerifyNow assay 2-4 h after all the antiplatelet agents are taken simultaneously in the morning at the end of Stage 1 (Visit 2) [ i.e., on the 4th (3rd-5th) week of treatment ]
Platelet reactivity index (PRI) | On the 12th (11th-13th) week of treatment
  The platelet reactivity index (PRI) assessed by vasodilator-stimulated phosphoprotein-phosphorylation (VASP-P) assay 2-4 h after all the antiplatelet agents are taken simultaneously in the morning at the end of the treatment period (Visit 4, EOT) [ i.e., on the 12th (11th-13th) week of treatment ]
Platelet reactivity index (PRI) | On the 8th (7th-9th) week of treatment
  The platelet reactivity index (PRI) assessed by vasodilator-stimulated phosphoprotein-phosphorylation (VASP-P) assay 2-4 h after all the antiplatelet agents are taken simultaneously in the morning at the end of Stage 2 (Visit 3) [ i.e., on the 8th (7th-9th) week of treatment ]
Platelet reactivity index (PRI) | On the 4th (3rd-5th) week of treatment
  The platelet reactivity index (PRI) assessed by vasodilator-stimulated phosphoprotein-phosphorylation (VASP-P) assay 2-4 h after all the antiplatelet agents are taken simultaneously in the morning at the end of Stage 1 (Visit 2) [ i.e., on the 4th (3rd-5th) week of treatment ]
Urinary 11-dehydro-thromboxane B2 (11-dH-TXB2) | On the 12th (11th-13th) week of treatment
  The urinary 11-dehydro-thromboxane B2 (11-dH-TXB2) assessed by enzyme-linked immunosorbent assay (ELISA) 2-4 h after all the antiplatelet agents are taken simultaneously in the morning at the end of the treatment period (Visit 4, EOT) [ i.e., on the 12th (11th-13th) week of treatment ]
Urinary 11-dehydro-thromboxane B2 (11-dH-TXB2) | On the 8th (7th-9th) week of treatment
  The urinary 11-dehydro-thromboxane B2 (11-dH-TXB2) assessed by enzyme-linked immunosorbent assay (ELISA) 2-4 h after all the antiplatelet agents are taken simultaneously in the morning at the end of Stage 2 (Visit 3) [ i.e., on the 8th (7th-9th) week of treatment ]
Urinary 11-dehydro-thromboxane B2 (11-dH-TXB2) | On the 4th (3rd-5th) week of treatment
  The urinary 11-dehydro-thromboxane B2 (11-dH-TXB2) assessed by enzyme-linked immunosorbent assay (ELISA) 2-4 h after all the antiplatelet agents are taken simultaneously in the morning at the end of Stage 1 (Visit 2) [ i.e., on the 4th (3rd-5th) week of treatment ]

OTHER OUTCOMES:
Major adverse cardiac events (MACE) | Up to the 12th (11th-13th) week of treatment
  The composite of death, or myocardial infarction, or urgent coronary revascularization, or definite or possible stent thrombosis, up to the end of the treatment period (Visit 4, EOT), i.e., the 12th (11th-13th) week of treatment
Major bleeding | Up to the 12th (11th-13th) week of treatment
  The major bleeding according to platelet inhibition and patient outcomes (PLATO) definition up to the end of the treatment period (Visit 4, EOT), i.e., the 12th (11th-13th) week of treatment
Minor bleeding | Up to the 12th (11th-13th) week of treatment
  The minor bleeding according to platelet inhibition and patient outcomes (PLATO) definition up to the end of the treatment period (Visit 4, EOT), i.e., the 12th (11th-13th) week of treatment
Minimal bleeding | Up to the 12th (11th-13th) week of treatment
  The minimal bleeding according to platelet inhibition and patient outcomes (PLATO) definition up to the end of the treatment period (Visit 4, EOT), i.e., the 12th (11th-13th) week of treatment
Major or minor bleeding | Up to the 12th (11th-13th) week of treatment
  The major or minor bleeding according to platelet inhibition and patient outcomes (PLATO) definition up to the end of the treatment period (Visit 4, EOT), i.e., the 12th (11th-13th) week of treatment
Major or minor or minimal bleeding | Up to the 12th (11th-13th) week of treatment
  The major or minor or minimal bleeding according to platelet inhibition and patient outcomes (PLATO) definition up to the end of the treatment period (Visit 4, EOT), i.e., the 12th (11th-13th) week of treatment
P-selectin (CD62p) expression | On the 12th (11th-13th) week of treatment
  The P-selectin (CD62p) expression assessed by flow cytometry 2-4 h after all the antiplatelet agents are taken simultaneously in the morning at the end of the treatment period (Visit 4, EOT) [ i.e., the 12th (11th-13th) week of treatment ]
Serum soluble P-selectin (sCD62p) | On the 12th (11th-13th) week of treatment
  Serum soluble P-selectin (sCD62p) assessed by enzyme-linked immunosorbent assay (ELISA) 2-4 h after all the antiplatelet agents are taken simultaneously in the morning at the end of the treatment period (Visit 4, EOT) [ i.e., on the 12th (11th-13th) week of treatment ]
Serum soluble CD40 ligand (sCD40L) | On the 12th (11th-13th) week of treatment
  Serum soluble CD40 ligand (sCD40L) assessed by enzyme-linked immunosorbent assay (ELISA) 2-4 h after all the antiplatelet agents are taken simultaneously in the morning at the end of the treatment period (Visit 4, EOT) [ i.e., on the 12th (11th-13th) week of treatment ]

CONTACTS AND LOCATIONS:
Overall Officials: Zhenyu Liu, M.D., Principal Investigator — Department of Cardiology, Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Amsterdam EA, Wenger NK, Brindis RG, Casey DE Jr, Ganiats TG, Holmes DR Jr, Jaffe AS, Jneid H, Kelly RF, Kontos MC, Levine GN, Liebson PR, Mukherjee D, Peterson ED, Sabatine MS, Smalling RW, Zieman SJ. 2014 AHA/ACC Guideline for the Management of Patients with Non-ST-Elevation Acute Coronary Syndromes: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines. J Am Coll Cardiol. 2014 Dec 23;64(24):e139-e228. doi: 10.1016/j.jacc.2014.09.017. Epub 2014 Sep 23. No abstract available. PMID 25260718
- [Background] Aradi D, Komocsi A, Vorobcsuk A, Rideg O, Tokes-Fuzesi M, Magyarlaki T, Horvath IG, Serebruany VL. Prognostic significance of high on-clopidogrel platelet reactivity after percutaneous coronary intervention: systematic review and meta-analysis. Am Heart J. 2010 Sep;160(3):543-51. doi: 10.1016/j.ahj.2010.06.004. PMID 20826265
- [Background] Aradi D, Storey RF, Komocsi A, Trenk D, Gulba D, Kiss RG, Husted S, Bonello L, Sibbing D, Collet JP, Huber K; Working Group on Thrombosis of the European Society of Cardiology. Expert position paper on the role of platelet function testing in patients undergoing percutaneous coronary intervention. Eur Heart J. 2014 Jan;35(4):209-15. doi: 10.1093/eurheartj/eht375. Epub 2013 Sep 25. No abstract available. PMID 24067509
- [Background] Bonaca MP, Bhatt DL, Cohen M, Steg PG, Storey RF, Jensen EC, Magnani G, Bansilal S, Fish MP, Im K, Bengtsson O, Oude Ophuis T, Budaj A, Theroux P, Ruda M, Hamm C, Goto S, Spinar J, Nicolau JC, Kiss RG, Murphy SA, Wiviott SD, Held P, Braunwald E, Sabatine MS; PEGASUS-TIMI 54 Steering Committee and Investigators. Long-term use of ticagrelor in patients with prior myocardial infarction. N Engl J Med. 2015 May 7;372(19):1791-800. doi: 10.1056/NEJMoa1500857. Epub 2015 Mar 14. PMID 25773268
- [Background] Bonello L, Camoin-Jau L, Arques S, Boyer C, Panagides D, Wittenberg O, Simeoni MC, Barragan P, Dignat-George F, Paganelli F. Adjusted clopidogrel loading doses according to vasodilator-stimulated phosphoprotein phosphorylation index decrease rate of major adverse cardiovascular events in patients with clopidogrel resistance: a multicenter randomized prospective study. J Am Coll Cardiol. 2008 Apr 8;51(14):1404-11. doi: 10.1016/j.jacc.2007.12.044. PMID 18387444
- [Background] Brar SS, ten Berg J, Marcucci R, Price MJ, Valgimigli M, Kim HS, Patti G, Breet NJ, DiSciascio G, Cuisset T, Dangas G. Impact of platelet reactivity on clinical outcomes after percutaneous coronary intervention. A collaborative meta-analysis of individual participant data. J Am Coll Cardiol. 2011 Nov 1;58(19):1945-54. doi: 10.1016/j.jacc.2011.06.059. PMID 22032704
- [Background] Caliceti C, Franco P, Spinozzi S, Roda A, Cicero AF. Berberine: New Insights from Pharmacological Aspects to Clinical Evidences in the Management of Metabolic Disorders. Curr Med Chem. 2016;23(14):1460-76. doi: 10.2174/0929867323666160411143314. PMID 27063256
- [Background] Chen JJ, Chang YL, Teng CM, Lin WY, Chen YC, Chen IS. A new tetrahydroprotoberberine N-oxide alkaloid and anti-platelet aggregation constituents of Corydalis tashiroi. Planta Med. 2001 Jul;67(5):423-7. doi: 10.1055/s-2001-15820. PMID 11488455
- [Background] Chu JW, Wong CK, Chambers J, Wout JV, Herbison P, Tang EW. Aspirin resistance determined from a bed-side test in patients suspected to have acute coronary syndrome portends a worse 6 months outcome. QJM. 2010 Jun;103(6):405-12. doi: 10.1093/qjmed/hcq038. Epub 2010 Mar 30. PMID 20356848
- [Background] Combescure C, Fontana P, Mallouk N, Berdague P, Labruyere C, Barazer I, Gris JC, Laporte S, Fabbro-Peray P, Reny JL; CLOpidogrel and Vascular ISchemic Events Meta-analysis Study Group. Clinical implications of clopidogrel non-response in cardiovascular patients: a systematic review and meta-analysis. J Thromb Haemost. 2010 May;8(5):923-33. doi: 10.1111/j.1538-7836.2010.03809.x. Epub 2010 Feb 12. PMID 20156305
- [Background] Fritsma GA, Ens GE, Alvord MA, Carroll AA, Jensen R. Monitoring the antiplatelet action of aspirin. JAAPA. 2001 May;14(5):57-8, 61-2. No abstract available. PMID 11523339
- [Background] Glauser J, Emerman CL, Bhatt DL, Peacock WF 4th. Platelet aspirin resistance in ED patients with suspected acute coronary syndrome. Am J Emerg Med. 2010 May;28(4):440-4. doi: 10.1016/j.ajem.2009.01.004. PMID 20466222
- [Background] Gurbel PA, Bliden KP, Butler K, Tantry US, Gesheff T, Wei C, Teng R, Antonino MJ, Patil SB, Karunakaran A, Kereiakes DJ, Parris C, Purdy D, Wilson V, Ledley GS, Storey RF. Randomized double-blind assessment of the ONSET and OFFSET of the antiplatelet effects of ticagrelor versus clopidogrel in patients with stable coronary artery disease: the ONSET/OFFSET study. Circulation. 2009 Dec 22;120(25):2577-85. doi: 10.1161/CIRCULATIONAHA.109.912550. Epub 2009 Nov 18. PMID 19923168
- [Background] Gurbel PA, Bliden KP, Butler K, Antonino MJ, Wei C, Teng R, Rasmussen L, Storey RF, Nielsen T, Eikelboom JW, Sabe-Affaki G, Husted S, Kereiakes DJ, Henderson D, Patel DV, Tantry US. Response to ticagrelor in clopidogrel nonresponders and responders and effect of switching therapies: the RESPOND study. Circulation. 2010 Mar 16;121(10):1188-99. doi: 10.1161/CIRCULATIONAHA.109.919456. Epub 2010 Mar 1. PMID 20194878
- [Background] Huang CG, Chu ZL, Wei SJ, Jiang H, Jiao BH. Effect of berberine on arachidonic acid metabolism in rabbit platelets and endothelial cells. Thromb Res. 2002 May 15;106(4-5):223-7. doi: 10.1016/s0049-3848(02)00133-0. PMID 12297129
- [Background] Husted S, Emanuelsson H, Heptinstall S, Sandset PM, Wickens M, Peters G. Pharmacodynamics, pharmacokinetics, and safety of the oral reversible P2Y12 antagonist AZD6140 with aspirin in patients with atherosclerosis: a double-blind comparison to clopidogrel with aspirin. Eur Heart J. 2006 May;27(9):1038-47. doi: 10.1093/eurheartj/ehi754. Epub 2006 Feb 13. PMID 16476694
- [Background] James S, Akerblom A, Cannon CP, Emanuelsson H, Husted S, Katus H, Skene A, Steg PG, Storey RF, Harrington R, Becker R, Wallentin L. Comparison of ticagrelor, the first reversible oral P2Y(12) receptor antagonist, with clopidogrel in patients with acute coronary syndromes: Rationale, design, and baseline characteristics of the PLATelet inhibition and patient Outcomes (PLATO) trial. Am Heart J. 2009 Apr;157(4):599-605. doi: 10.1016/j.ahj.2009.01.003. PMID 19332184
- [Background] Kamath S, Blann AD, Lip GY. Platelet activation: assessment and quantification. Eur Heart J. 2001 Sep;22(17):1561-71. doi: 10.1053/euhj.2000.2515. No abstract available. PMID 11492985
- [Background] Lan J, Zhao Y, Dong F, Yan Z, Zheng W, Fan J, Sun G. Meta-analysis of the effect and safety of berberine in the treatment of type 2 diabetes mellitus, hyperlipemia and hypertension. J Ethnopharmacol. 2015 Feb 23;161:69-81. doi: 10.1016/j.jep.2014.09.049. Epub 2014 Dec 10. PMID 25498346
- [Background] Levine GN, Bates ER, Blankenship JC, Bailey SR, Bittl JA, Cercek B, Chambers CE, Ellis SG, Guyton RA, Hollenberg SM, Khot UN, Lange RA, Mauri L, Mehran R, Moussa ID, Mukherjee D, Nallamothu BK, Ting HH; American College of Cardiology Foundation; American Heart Association Task Force on Practice Guidelines; Society for Cardiovascular Angiography and Interventions. 2011 ACCF/AHA/SCAI Guideline for Percutaneous Coronary Intervention. A report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines and the Society for Cardiovascular Angiography and Interventions. J Am Coll Cardiol. 2011 Dec 6;58(24):e44-122. doi: 10.1016/j.jacc.2011.08.007. Epub 2011 Nov 7. No abstract available. PMID 22070834
- [Background] Levine GN, Bates ER, Bittl JA, Brindis RG, Fihn SD, Fleisher LA, Granger CB, Lange RA, Mack MJ, Mauri L, Mehran R, Mukherjee D, Newby LK, O'Gara PT, Sabatine MS, Smith PK, Smith SC Jr. 2016 ACC/AHA Guideline Focused Update on Duration of Dual Antiplatelet Therapy in Patients With Coronary Artery Disease: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. J Am Coll Cardiol. 2016 Sep 6;68(10):1082-115. doi: 10.1016/j.jacc.2016.03.513. Epub 2016 Mar 29. No abstract available. PMID 27036918
- [Background] Lordkipanidze M, Pharand C, Schampaert E, Turgeon J, Palisaitis DA, Diodati JG. A comparison of six major platelet function tests to determine the prevalence of aspirin resistance in patients with stable coronary artery disease. Eur Heart J. 2007 Jul;28(14):1702-8. doi: 10.1093/eurheartj/ehm226. Epub 2007 Jun 14. PMID 17569678
- [Background] Malinin A, Pokov A, Spergling M, Defranco A, Schwartz K, Schwartz D, Mahmud E, Atar D, Serebruany V. Monitoring platelet inhibition after clopidogrel with the VerifyNow-P2Y12(R) rapid analyzer: the VERIfy Thrombosis risk ASsessment (VERITAS) study. Thromb Res. 2007;119(3):277-84. doi: 10.1016/j.thromres.2006.01.019. Epub 2006 Mar 24. PMID 16563469
- [Background] Mauri L, Hsieh WH, Massaro JM, Ho KK, D'Agostino R, Cutlip DE. Stent thrombosis in randomized clinical trials of drug-eluting stents. N Engl J Med. 2007 Mar 8;356(10):1020-9. doi: 10.1056/NEJMoa067731. Epub 2007 Feb 12. PMID 17296821
- [Background] CURRENT-OASIS 7 Investigators; Mehta SR, Bassand JP, Chrolavicius S, Diaz R, Eikelboom JW, Fox KA, Granger CB, Jolly S, Joyner CD, Rupprecht HJ, Widimsky P, Afzal R, Pogue J, Yusuf S. Dose comparisons of clopidogrel and aspirin in acute coronary syndromes. N Engl J Med. 2010 Sep 2;363(10):930-42. doi: 10.1056/NEJMoa0909475. PMID 20818903
- [Background] Mehta SR, Tanguay JF, Eikelboom JW, Jolly SS, Joyner CD, Granger CB, Faxon DP, Rupprecht HJ, Budaj A, Avezum A, Widimsky P, Steg PG, Bassand JP, Montalescot G, Macaya C, Di Pasquale G, Niemela K, Ajani AE, White HD, Chrolavicius S, Gao P, Fox KA, Yusuf S; CURRENT-OASIS 7 trial investigators. Double-dose versus standard-dose clopidogrel and high-dose versus low-dose aspirin in individuals undergoing percutaneous coronary intervention for acute coronary syndromes (CURRENT-OASIS 7): a randomised factorial trial. Lancet. 2010 Oct 9;376(9748):1233-43. doi: 10.1016/S0140-6736(10)61088-4. PMID 20817281
- [Background] Meng S, Wang LS, Huang ZQ, Zhou Q, Sun YG, Cao JT, Li YG, Wang CQ. Berberine ameliorates inflammation in patients with acute coronary syndrome following percutaneous coronary intervention. Clin Exp Pharmacol Physiol. 2012 May;39(5):406-11. doi: 10.1111/j.1440-1681.2012.05670.x. PMID 22220931
- [Background] Task Force Members; Montalescot G, Sechtem U, Achenbach S, Andreotti F, Arden C, Budaj A, Bugiardini R, Crea F, Cuisset T, Di Mario C, Ferreira JR, Gersh BJ, Gitt AK, Hulot JS, Marx N, Opie LH, Pfisterer M, Prescott E, Ruschitzka F, Sabate M, Senior R, Taggart DP, van der Wall EE, Vrints CJ; ESC Committee for Practice Guidelines; Zamorano JL, Achenbach S, Baumgartner H, Bax JJ, Bueno H, Dean V, Deaton C, Erol C, Fagard R, Ferrari R, Hasdai D, Hoes AW, Kirchhof P, Knuuti J, Kolh P, Lancellotti P, Linhart A, Nihoyannopoulos P, Piepoli MF, Ponikowski P, Sirnes PA, Tamargo JL, Tendera M, Torbicki A, Wijns W, Windecker S; Document Reviewers; Knuuti J, Valgimigli M, Bueno H, Claeys MJ, Donner-Banzhoff N, Erol C, Frank H, Funck-Brentano C, Gaemperli O, Gonzalez-Juanatey JR, Hamilos M, Hasdai D, Husted S, James SK, Kervinen K, Kolh P, Kristensen SD, Lancellotti P, Maggioni AP, Piepoli MF, Pries AR, Romeo F, Ryden L, Simoons ML, Sirnes PA, Steg PG, Timmis A, Wijns W, Windecker S, Yildirir A, Zamorano JL. 2013 ESC guidelines on the management of stable coronary artery disease: the Task Force on the management of stable coronary artery disease of the European Society of Cardiology. Eur Heart J. 2013 Oct;34(38):2949-3003. doi: 10.1093/eurheartj/eht296. Epub 2013 Aug 30. No abstract available. PMID 23996286
- [Background] Montalescot G, van 't Hof AW, Lapostolle F, Silvain J, Lassen JF, Bolognese L, Cantor WJ, Cequier A, Chettibi M, Goodman SG, Hammett CJ, Huber K, Janzon M, Merkely B, Storey RF, Zeymer U, Stibbe O, Ecollan P, Heutz WM, Swahn E, Collet JP, Willems FF, Baradat C, Licour M, Tsatsaris A, Vicaut E, Hamm CW; ATLANTIC Investigators. Prehospital ticagrelor in ST-segment elevation myocardial infarction. N Engl J Med. 2014 Sep 11;371(11):1016-27. doi: 10.1056/NEJMoa1407024. Epub 2014 Sep 1. PMID 25175921
- [Background] O'Gara PT, Kushner FG, Ascheim DD, Casey DE Jr, Chung MK, de Lemos JA, Ettinger SM, Fang JC, Fesmire FM, Franklin BA, Granger CB, Krumholz HM, Linderbaum JA, Morrow DA, Newby LK, Ornato JP, Ou N, Radford MJ, Tamis-Holland JE, Tommaso CL, Tracy CM, Woo YJ, Zhao DX. 2013 ACCF/AHA guideline for the management of ST-elevation myocardial infarction: a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines. J Am Coll Cardiol. 2013 Jan 29;61(4):e78-e140. doi: 10.1016/j.jacc.2012.11.019. Epub 2012 Dec 17. No abstract available. PMID 23256914
- [Background] Pang B, Zhao LH, Zhou Q, Zhao TY, Wang H, Gu CJ, Tong XL. Application of berberine on treating type 2 diabetes mellitus. Int J Endocrinol. 2015;2015:905749. doi: 10.1155/2015/905749. Epub 2015 Mar 11. PMID 25861268
- [Background] Perneby C, Granstrom E, Beck O, Fitzgerald D, Harhen B, Hjemdahl P. Optimization of an enzyme immunoassay for 11-dehydro-thromboxane B(2) in urine: comparison with GC-MS. Thromb Res. 1999 Dec 15;96(6):427-36. doi: 10.1016/s0049-3848(99)00126-7. PMID 10632465
- [Background] Pirillo A, Catapano AL. Berberine, a plant alkaloid with lipid- and glucose-lowering properties: From in vitro evidence to clinical studies. Atherosclerosis. 2015 Dec;243(2):449-61. doi: 10.1016/j.atherosclerosis.2015.09.032. Epub 2015 Sep 30. PMID 26520899
- [Background] Price MJ, Endemann S, Gollapudi RR, Valencia R, Stinis CT, Levisay JP, Ernst A, Sawhney NS, Schatz RA, Teirstein PS. Prognostic significance of post-clopidogrel platelet reactivity assessed by a point-of-care assay on thrombotic events after drug-eluting stent implantation. Eur Heart J. 2008 Apr;29(8):992-1000. doi: 10.1093/eurheartj/ehn046. Epub 2008 Feb 10. PMID 18263931
- [Background] Price MJ, Berger PB, Teirstein PS, Tanguay JF, Angiolillo DJ, Spriggs D, Puri S, Robbins M, Garratt KN, Bertrand OF, Stillabower ME, Aragon JR, Kandzari DE, Stinis CT, Lee MS, Manoukian SV, Cannon CP, Schork NJ, Topol EJ; GRAVITAS Investigators. Standard- vs high-dose clopidogrel based on platelet function testing after percutaneous coronary intervention: the GRAVITAS randomized trial. JAMA. 2011 Mar 16;305(11):1097-105. doi: 10.1001/jama.2011.290. PMID 21406646
- [Background] Ramstrom S, Sodergren AL, Tynngard N, Lindahl TL. Platelet Function Determined by Flow Cytometry: New Perspectives? Semin Thromb Hemost. 2016 Apr;42(3):268-81. doi: 10.1055/s-0035-1570082. Epub 2016 Feb 17. PMID 26886398
- [Background] Roffi M, Patrono C, Collet JP, Mueller C, Valgimigli M, Andreotti F, Bax JJ, Borger MA, Brotons C, Chew DP, Gencer B, Hasenfuss G, Kjeldsen K, Lancellotti P, Landmesser U, Mehilli J, Mukherjee D, Storey RF, Windecker S; ESC Scientific Document Group. 2015 ESC Guidelines for the management of acute coronary syndromes in patients presenting without persistent ST-segment elevation: Task Force for the Management of Acute Coronary Syndromes in Patients Presenting without Persistent ST-Segment Elevation of the European Society of Cardiology (ESC). Eur Heart J. 2016 Jan 14;37(3):267-315. doi: 10.1093/eurheartj/ehv320. Epub 2015 Aug 29. No abstract available. PMID 26320110
- [Background] Rubak P, Nissen PH, Kristensen SD, Hvas AM. Investigation of platelet function and platelet disorders using flow cytometry. Platelets. 2016;27(1):66-74. doi: 10.3109/09537104.2015.1032919. Epub 2015 Apr 22. PMID 25901600
- [Background] Schwarz UR, Geiger J, Walter U, Eigenthaler M. Flow cytometry analysis of intracellular VASP phosphorylation for the assessment of activating and inhibitory signal transduction pathways in human platelets--definition and detection of ticlopidine/clopidogrel effects. Thromb Haemost. 1999 Sep;82(3):1145-52. PMID 10494779
- [Background] Shah BH, Nawaz Z, Saeed SA. Gilani AH. Agonist-dependent Differential Effects of Berberine in Human Platelet Aggregation. Phytother. Res. 12, S60-S62 (1998).
- [Background] Sofi F, Marcucci R, Gori AM, Giusti B, Abbate R, Gensini GF. Clopidogrel non-responsiveness and risk of cardiovascular morbidity. An updated meta-analysis. Thromb Haemost. 2010 Apr;103(4):841-8. doi: 10.1160/TH09-06-0418. Epub 2010 Feb 2. PMID 20135063
- [Background] Task Force on the management of ST-segment elevation acute myocardial infarction of the European Society of Cardiology (ESC); Steg PG, James SK, Atar D, Badano LP, Blomstrom-Lundqvist C, Borger MA, Di Mario C, Dickstein K, Ducrocq G, Fernandez-Aviles F, Gershlick AH, Giannuzzi P, Halvorsen S, Huber K, Juni P, Kastrati A, Knuuti J, Lenzen MJ, Mahaffey KW, Valgimigli M, van 't Hof A, Widimsky P, Zahger D. ESC Guidelines for the management of acute myocardial infarction in patients presenting with ST-segment elevation. Eur Heart J. 2012 Oct;33(20):2569-619. doi: 10.1093/eurheartj/ehs215. Epub 2012 Aug 24. No abstract available. PMID 22922416
- [Background] Stone GW, Witzenbichler B, Weisz G, Rinaldi MJ, Neumann FJ, Metzger DC, Henry TD, Cox DA, Duffy PL, Mazzaferri E, Gurbel PA, Xu K, Parise H, Kirtane AJ, Brodie BR, Mehran R, Stuckey TD; ADAPT-DES Investigators. Platelet reactivity and clinical outcomes after coronary artery implantation of drug-eluting stents (ADAPT-DES): a prospective multicentre registry study. Lancet. 2013 Aug 17;382(9892):614-23. doi: 10.1016/S0140-6736(13)61170-8. Epub 2013 Jul 26. PMID 23890998
- [Background] Storey RF, Husted S, Harrington RA, Heptinstall S, Wilcox RG, Peters G, Wickens M, Emanuelsson H, Gurbel P, Grande P, Cannon CP. Inhibition of platelet aggregation by AZD6140, a reversible oral P2Y12 receptor antagonist, compared with clopidogrel in patients with acute coronary syndromes. J Am Coll Cardiol. 2007 Nov 6;50(19):1852-6. doi: 10.1016/j.jacc.2007.07.058. Epub 2007 Oct 23. PMID 17980251
- [Background] Storey RF, Angiolillo DJ, Patil SB, Desai B, Ecob R, Husted S, Emanuelsson H, Cannon CP, Becker RC, Wallentin L. Inhibitory effects of ticagrelor compared with clopidogrel on platelet function in patients with acute coronary syndromes: the PLATO (PLATelet inhibition and patient Outcomes) PLATELET substudy. J Am Coll Cardiol. 2010 Oct 26;56(18):1456-62. doi: 10.1016/j.jacc.2010.03.100. PMID 20832963
- [Background] Tantry US, Bonello L, Aradi D, Price MJ, Jeong YH, Angiolillo DJ, Stone GW, Curzen N, Geisler T, Ten Berg J, Kirtane A, Siller-Matula J, Mahla E, Becker RC, Bhatt DL, Waksman R, Rao SV, Alexopoulos D, Marcucci R, Reny JL, Trenk D, Sibbing D, Gurbel PA; Working Group on On-Treatment Platelet Reactivity. Consensus and update on the definition of on-treatment platelet reactivity to adenosine diphosphate associated with ischemia and bleeding. J Am Coll Cardiol. 2013 Dec 17;62(24):2261-73. doi: 10.1016/j.jacc.2013.07.101. Epub 2013 Sep 27. PMID 24076493
- [Background] Thygesen K, Alpert JS, Jaffe AS, Simoons ML, Chaitman BR, White HD; Writing Group on the Joint ESC/ACCF/AHA/WHF Task Force for the Universal Definition of Myocardial Infarction; Thygesen K, Alpert JS, White HD, Jaffe AS, Katus HA, Apple FS, Lindahl B, Morrow DA, Chaitman BA, Clemmensen PM, Johanson P, Hod H, Underwood R, Bax JJ, Bonow RO, Pinto F, Gibbons RJ, Fox KA, Atar D, Newby LK, Galvani M, Hamm CW, Uretsky BF, Steg PG, Wijns W, Bassand JP, Menasche P, Ravkilde J, Ohman EM, Antman EM, Wallentin LC, Armstrong PW, Simoons ML, Januzzi JL, Nieminen MS, Gheorghiade M, Filippatos G, Luepker RV, Fortmann SP, Rosamond WD, Levy D, Wood D, Smith SC, Hu D, Lopez-Sendon JL, Robertson RM, Weaver D, Tendera M, Bove AA, Parkhomenko AN, Vasilieva EJ, Mendis S; ESC Committee for Practice Guidelines (CPG). Third universal definition of myocardial infarction. Eur Heart J. 2012 Oct;33(20):2551-67. doi: 10.1093/eurheartj/ehs184. Epub 2012 Aug 24. No abstract available. PMID 22922414
- [Background] van Velzen JF, Laros-van Gorkom BA, Pop GA, van Heerde WL. Multicolor flow cytometry for evaluation of platelet surface antigens and activation markers. Thromb Res. 2012 Jul;130(1):92-8. doi: 10.1016/j.thromres.2012.02.041. Epub 2012 Mar 16. PMID 22424855
- [Background] Wallentin L, Becker RC, Budaj A, Cannon CP, Emanuelsson H, Held C, Horrow J, Husted S, James S, Katus H, Mahaffey KW, Scirica BM, Skene A, Steg PG, Storey RF, Harrington RA; PLATO Investigators; Freij A, Thorsen M. Ticagrelor versus clopidogrel in patients with acute coronary syndromes. N Engl J Med. 2009 Sep 10;361(11):1045-57. doi: 10.1056/NEJMoa0904327. Epub 2009 Aug 30. PMID 19717846
- [Background] Authors/Task Force members; Windecker S, Kolh P, Alfonso F, Collet JP, Cremer J, Falk V, Filippatos G, Hamm C, Head SJ, Juni P, Kappetein AP, Kastrati A, Knuuti J, Landmesser U, Laufer G, Neumann FJ, Richter DJ, Schauerte P, Sousa Uva M, Stefanini GG, Taggart DP, Torracca L, Valgimigli M, Wijns W, Witkowski A. 2014 ESC/EACTS Guidelines on myocardial revascularization: The Task Force on Myocardial Revascularization of the European Society of Cardiology (ESC) and the European Association for Cardio-Thoracic Surgery (EACTS)Developed with the special contribution of the European Association of Percutaneous Cardiovascular Interventions (EAPCI). Eur Heart J. 2014 Oct 1;35(37):2541-619. doi: 10.1093/eurheartj/ehu278. Epub 2014 Aug 29. No abstract available. PMID 25173339
- [Background] Wiviott SD, Braunwald E, McCabe CH, Montalescot G, Ruzyllo W, Gottlieb S, Neumann FJ, Ardissino D, De Servi S, Murphy SA, Riesmeyer J, Weerakkody G, Gibson CM, Antman EM; TRITON-TIMI 38 Investigators. Prasugrel versus clopidogrel in patients with acute coronary syndromes. N Engl J Med. 2007 Nov 15;357(20):2001-15. doi: 10.1056/NEJMoa0706482. Epub 2007 Nov 4. PMID 17982182
- [Background] Wiviott SD, Trenk D, Frelinger AL, O'Donoghue M, Neumann FJ, Michelson AD, Angiolillo DJ, Hod H, Montalescot G, Miller DL, Jakubowski JA, Cairns R, Murphy SA, McCabe CH, Antman EM, Braunwald E; PRINCIPLE-TIMI 44 Investigators. Prasugrel compared with high loading- and maintenance-dose clopidogrel in patients with planned percutaneous coronary intervention: the Prasugrel in Comparison to Clopidogrel for Inhibition of Platelet Activation and Aggregation-Thrombolysis in Myocardial Infarction 44 trial. Circulation. 2007 Dec 18;116(25):2923-32. doi: 10.1161/CIRCULATIONAHA.107.740324. Epub 2007 Dec 3. PMID 18056526
- [Background] Yu J, Mehran R, Dangas GD, Claessen BE, Baber U, Xu K, Parise H, Fahy M, Lansky AJ, Witzenbichler B, Grines CL, Guagliumi G, Kornowski R, Wohrle J, Dudek D, Weisz G, Stone GW. Safety and efficacy of high- versus low-dose aspirin after primary percutaneous coronary intervention in ST-segment elevation myocardial infarction: the HORIZONS-AMI (Harmonizing Outcomes With Revascularization and Stents in Acute Myocardial Infarction) trial. JACC Cardiovasc Interv. 2012 Dec;5(12):1231-8. doi: 10.1016/j.jcin.2012.07.016. PMID 23257371
- [Background] Yun SH, Sim EH, Goh RY, Park JI, Han JY. Platelet Activation: The Mechanisms and Potential Biomarkers. Biomed Res Int. 2016;2016:9060143. doi: 10.1155/2016/9060143. Epub 2016 Jun 15. PMID 27403440
- [Background] Yusuf S, Zhao F, Mehta SR, Chrolavicius S, Tognoni G, Fox KK; Clopidogrel in Unstable Angina to Prevent Recurrent Events Trial Investigators. Effects of clopidogrel in addition to aspirin in patients with acute coronary syndromes without ST-segment elevation. N Engl J Med. 2001 Aug 16;345(7):494-502. doi: 10.1056/NEJMoa010746. PMID 11519503
- [Background] Zhang Y, Ma XJ, Guo CY, Wang MM, Kou N, Qu H, Mao HM, Shi DZ. Pretreatment with a combination of ligustrazine and berberine improves cardiac function in rats with coronary microembolization. Acta Pharmacol Sin. 2016 Apr;37(4):463-72. doi: 10.1038/aps.2015.147. Epub 2016 Feb 29. PMID 26924290